CLINICAL TRIAL: NCT02690207
Title: Cross-vaccination Study of GSK Biologicals' Lyophilized Formulation of the Herpes Zoster Subunit (HZ/su) Vaccine (GSK 1437173A) in Subjects Who Previously Received Placebo in ZOSTER-006 (NCT01165177) and ZOSTER-022 (NCT01165229) Studies
Brief Title: Cross-vaccination Study of GSK Biologicals' Herpes Zoster Subunit (HZ/su) Vaccine (GSK 1437173A) in Subjects Who Previously Received Placebo in ZOSTER-006 (NCT01165177) and ZOSTER-022 (NCT01165229) Studies.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 204486; 2015-000965-30 (EudraCT Number)
Record Dates: First submitted 2016-02-16; First posted 2016-02-24 (Estimated); Results first posted 2020-03-12 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-02

CONDITIONS: Herpes Zoster
Keywords: Herpes Zoster; Safety; Adults; Cross-vaccination
MeSH Terms: conditions — Herpes Zoster

ARMS (1):
- HZ/su Group (Experimental): Subjects received Herpes Zoster subunit vaccine, administered intramuscularly (IM) in the deltoid of the non-dominant arm
  Interventions: Biological: Herpes Zoster Vaccine GSK1437173A

INTERVENTIONS:
Biological: Herpes Zoster Vaccine GSK1437173A — Intramuscular injection
  Other Names: HZ/su

SUMMARY:
The purpose of this study is to cross-vaccinate and collect safety data in terms of unsolicited Adverse Events (AEs), Serious Adverse Events (SAEs) and potential Immune Mediated Disease (pIMD) from subjects >= 50 Years of age (YOA) who previously received placebo in ZOSTER-006 (NCT01165177) and ZOSTER-022 (NCT01165229).

DETAILED DESCRIPTION:
Since the HZ/su vaccine has not yet been licensed and marketed, this study is being conducted to enable potentially eligible subjects who previously received placebo in ZOSTER-006 (NCT01165177) or ZOSTER-022 (NCT01165229) to receive the HZ/su vaccine.

Study ZOSTER-056 is an open-label, multi-centric and single arm study to cross-vaccinate and collect safety data in terms of of unsolicited Adverse Events (AEs), Serious Adverse Events (SAEs) and pIMD from subjects >= 50 YOA who previously received placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g. completion of the diary cards, vaccination visits, follow-up contacts). Or subjects' Legally Acceptable Representative(s) [LAR(s)]/caregiver who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g. completion of the diary cards, vaccination visits, availability for follow-up contacts).
* Written informed consent obtained from the subject/Legally Acceptable representative(s) [LAR(s)] of the subject prior to performing any study specific procedure. If the subjects is not capable of giving consent, his/her assent to participate should be obtained to the extent possible.
* Subject who previously participated in ZOSTER-006 or ZOSTER-022 studies and received at least one dose of placebo.
* Female subjects of non-childbearing potential may be enrolled in the study.

  * Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination and
  * has agreed to continue adequate contraception during the entire treatment period* and for 2 months after completion of the vaccination series.

    * treatment period refers to vaccination days and the interval between them.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine during the period starting 30 days before the first dose of study vaccine (Day -29 to Day 0), or planned use up to 30 days post Dose 2.
* Previous vaccination against Varicella Zoster virus (VZV) or HZ.
* Planned administration of VZV or HZ vaccination during the study (including an investigational or non-registered vaccine), with the exception of the study vaccine.
* Planned administration/administration of a vaccine/product not foreseen by the study protocol in the period starting 30 days before the first dose and ending 30 days after the last dose of vaccine administration, with the exception of licensed non-replicating vaccines (i.e. inactivated and subunit vaccines, including inactivated and subunit influenza vaccines, with or without adjuvant for seasonal or pandemic flus). These may be administered up to 8 days prior to dose 1 and/or dose 2 and/or at least 14 days after any dose of study vaccine
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting six months prior to the first vaccine dose and up to 30 days post Dose 2. For corticosteroids, this will mean prednisone ≥ 20 mg/day or equivalent. Inhaled, topical and intra-articular corticosteroids are allowed.
* Administration of long-acting immune-modifying drugs (e.g. infliximab, rituximab) within six months prior to the first vaccine dose up to 30 days post Dose 2.
* Concurrently participating in another clinical study, at the time of enrolment or planned participation up to the 30 days post second dose, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product (pharmaceutical product or device).
* Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease (e.g., malignancy, Human Immunodeficiency Virus [HIV] infection) or immunosuppressive/cytotoxic therapy (e.g., medications used during cancer chemotherapy, organ transplantation or to treat autoimmune disorders).
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Active HZ infection at the time of enrolment (i.e. HZ lesions not completely crusted over).
* Pregnant or lactating female.
* Any condition which, in the opinion of the investigator, prevents the subject from participating in the study.
* Any condition which in the judgment of the investigator would make intramuscular injection unsafe.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8687 (Actual)
Dates: Start 2016-03-16 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (169):
- United States (34):
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Spring Valley, California
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Meridian, Idaho
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Columbia, Maryland
  - GSK Investigational Site, Elkridge, Maryland
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Somers Point, New Jersey
  - GSK Investigational Site, Cary, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Hickory, North Carolina
  - GSK Investigational Site, Salisbury, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Wadsworth, Ohio
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Uniontown, Pennsylvania
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Murray, Utah
  - GSK Investigational Site, Newport News, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Winchester, Virginia
  - GSK Investigational Site, Renton, Washington
- Australia (7):
  - GSK Investigational Site, Maroubra, New South Wales
  - GSK Investigational Site, Umina, New South Wales
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Wollongong, New South Wales
  - GSK Investigational Site, Kippa-Ring, Queensland
  - GSK Investigational Site, Geelong, Victoria
  - GSK Investigational Site, Ivanhoe, Victoria
- Brazil (5):
  - GSK Investigational Site, Belo Horizonte, Minas Gerais
  - GSK Investigational Site, Curitiba, Paraná
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Curitiba/PR
  - GSK Investigational Site, São Paulo
- Canada (13):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Victoria, British Columbia
  - GSK Investigational Site, Bay Roberts, Newfoundland and Labrador
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Woodstock, Ontario
  - GSK Investigational Site, Gatineau, Quebec
  - GSK Investigational Site, Mirabel, Quebec
  - GSK Investigational Site, Pointe-Claire, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec
- Czechia (3):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, České Budějovice
  - GSK Investigational Site, Hradec Králové
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Finland (9):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Kokkola
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- France (12):
  - GSK Investigational Site, Angers
  - GSK Investigational Site, Château-Gontier
  - GSK Investigational Site, Clermont-Ferrand
  - GSK Investigational Site, Laval
  - GSK Investigational Site, Montrevault
  - GSK Investigational Site, Muret
  - GSK Investigational Site, Mûrs-Erigné
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Rosiers-d'Égletons
  - GSK Investigational Site, Saint-Cyr-sur-Loire
  - GSK Investigational Site, Segré
  - GSK Investigational Site, Tours
- Germany (28):
  - GSK Investigational Site, Deggingen, Baden-Wurttemberg
  - GSK Investigational Site, Güglingen, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Wangen, Baden-Wurttemberg
  - GSK Investigational Site, Weinheim, Baden-Wurttemberg
  - GSK Investigational Site, Dachau, Bavaria
  - GSK Investigational Site, Künzing, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Rednitzhembach, Bavaria
  - GSK Investigational Site, Wallerfing, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Flörsheim, Hesse
  - GSK Investigational Site, Duelmen, Lower Saxony
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Witten, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Rhaunen, Rhineland-Palatinate
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Freiberg, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Köthen, Saxony-Anhalt
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Magdeburg
- Hong Kong (2):
  - GSK Investigational Site, Kwun Tong
  - GSK Investigational Site, Shatin
- Italy (8):
  - GSK Investigational Site, Chieti, Abruzzo
  - GSK Investigational Site, Pescara, Abruzzo
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Monza, Lombardy
  - GSK Investigational Site, Cuneo, Piedmont
  - GSK Investigational Site, Sassari, Sardinia
  - GSK Investigational Site, Ragusa (RG), Sicily
- Japan (3):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Tokyo
- Mexico (4):
  - GSK Investigational Site, Zapopan, Jalisco, Jalisco
  - GSK Investigational Site, Jojutla, Morelos
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, Durango
- South Korea (6):
  - GSK Investigational Site, Ansan
  - GSK Investigational Site, Bucheon-si
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Kangnam-gu, Seoul
  - GSK Investigational Site, Kangwon-do
  - GSK Investigational Site, Seoul
- Spain (10):
  - GSK Investigational Site, Alcover( Tarragona)
  - GSK Investigational Site, Balenyà (Barcelona)
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Centelles (Barcelona)
  - GSK Investigational Site, La Roca Del Valles (Barcelona)
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Majadahonda( Madrid
  - GSK Investigational Site, Peralada( Girona)
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Vic
- Sweden (12):
  - GSK Investigational Site, Borås
  - GSK Investigational Site, Eskilstuna
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Jönköping
  - GSK Investigational Site, Karlskrona
  - GSK Investigational Site, Linköping
  - GSK Investigational Site, Malmo
  - GSK Investigational Site, Örebro
  - GSK Investigational Site, Skövde
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Uppsala
  - GSK Investigational Site, Vällingby
- Taiwan (3):
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan District
- United Kingdom (8):
  - GSK Investigational Site, Buckshaw Village, Chorley, Lancashire
  - GSK Investigational Site, Atherstone, Warwickshire
  - GSK Investigational Site, Bradford-on-Avon, Wiltshire
  - GSK Investigational Site, Bangor
  - GSK Investigational Site, Belfast
  - GSK Investigational Site, Broughshane
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, Newtonabbey

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20772

REFERENCES:
- [Background] Ocran-Appiah J, Boutry C, Herve C, Soni J, Schuind A; ZOSTER-056 Study Group. Safety of the adjuvanted recombinant zoster vaccine in adults aged 50 years or older. A phase IIIB, non-randomized, multinational, open-label study in previous ZOE-50 and ZOE-70 placebo recipients. Vaccine. 2021 Jan 3;39(1):6-10. doi: 10.1016/j.vaccine.2020.10.029. Epub 2020 Dec 1. PMID 33277059

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potentially eligible subjects who received placebo in ZOSTER-006 (NCT01165177) and ZOSTER-022 (NCT01165229) studies were enrolled in this study.
Pre-assignment Details: 8687 subjects were enrolled in this study and received Herpes Zoster sub-unit vaccine. Of these, 8434 subjects completed the trial and 253 subjects withdrew.
Period: Overall Study
Arm/Group | HZ/su Group
Started | 8687
Completed | 8434
Not Completed | 253
Not completed — Lost to Follow-up | 48
Not completed — Withdrawal by Subject | 46
Not completed — Protocol Violation | 2
Not completed — Serious adverse event | 110
Not completed — Non-serious Adverse Event | 18
Not completed — Migrated/moved from study area | 5
Not completed — Suspected HZ Episode | 1
Not completed — Other reasons for withdrawal | 23

BASELINE CHARACTERISTICS:
Arm/Group | HZ/su Group
Number analyzed (Participants) | 8687
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.6 (9.4)
Age, Customized [Count of Participants; unit: Participants]
  Age 18-64 years | 2326
  Age 65-84 years | 5574
  Age 85 years and over | 787
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 5254
  Male | 3433
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African Heritage/ African American | 72
  American Indian or Alaskan Native | 7
  Asian-Central/South Asian Heritage | 5
  Asian-East Asian Heritage | 1202
  Asian-Japanese Heritage | 254
  Asian-South East Asian Heritage | 12
  Native Hawaiian or Other Pacific Islander | 3
  White-Arabic/North African Heritage | 47
  White-Caucasian / European Heritage | 6361
  Other | 724

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related=AE assessed by the investigator as related to the vaccination.
Time Frame: During 30 days (Days 0-29) after any vaccination (across doses)
Population: This analysis was performed on Total vaccinated cohort, which included all subjects with at least one HZ/su vaccine administration documented for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | HZ/su Group
Number analyzed (Participants) | 8687
Participants
  Any AE(s) | 5175
  Grade 3 AE(s) | 963
  Related AE(s) | 4422

2. Primary Outcome: Number of Subjects With Any and Related Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that resulted in death, were life-threatening, required hospitalization or prolongation of hospitalization or resulted in disability/incapacity. Related=SAE assessed by the investigator as related to the vaccination.
Time Frame: From Month 0 until study end (Month 14, i.e. 12 months post dose 2)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HZ/su Group
Number analyzed (Participants) | 8687
Participants
  Any SAE(s) | 734
  Related SAE(s) | 2

3. Primary Outcome: Number of Subjects With Any and Related Potential Immune Mediated Diseases (pIMDs)
Description: pIMDs are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology. Related pIMDs=pIMDs assessed by the investigator as related to the vaccination.
Time Frame: From Month 0 until study end (Month 14, i.e. 12 months post dose 2)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HZ/su Group
Number analyzed (Participants) | 8687
Participants
  Any pIMD(s) | 62
  Related pIMD(s) | 1

4. Secondary Outcome: Number of Subjects With at Least One Suspected Herpes Zoster (HZ) Case(s)
Description: A suspected case of HZ was defined as a new rash characteristic of HZ (e.g., unilateral, dermatomal and accompanied by pain broadly defined to include allodynia, pruritus or other sensations).
  Clinically confirmed HZ episode is suspected HZ episode confirmed by the Investigator/Delegate.
Time Frame: From Month 0 until study end (Month 14, i.e. 12 months post dose 2)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HZ/su Group
Number analyzed (Participants) | 8687
Participants
  HZ episode | 30
  Suspected HZ episode only | 8
  Clinically confirmed HZ episode | 22

ADVERSE EVENTS:
Time Frame: Unsolicited AEs were collected during the 30 days (Days 0-29) follow-up period after any vaccination (across doses). SAEs were collected from Month 0 until study end (Month 14, i.e. 12 months post dose 2).
Arm/Group | HZ/su Group
All-Cause Mortality (participants affected / at risk) | 107/8687
Serious Adverse Events (participants affected / at risk) | 734/8687
Other Adverse Events (participants affected / at risk) | 5101/8687
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HZ/su Group (N=8687)
Anaemia (Blood and lymphatic system disorders) | 5 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 18 (19)
Angina pectoris (Cardiac disorders) | 12 (12)
Aortic valve stenosis (Cardiac disorders) | 2 (2)
Arrhythmia (Cardiac disorders) | 2 (2)
Arteriosclerosis coronary artery (Cardiac disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 25 (27)
Atrial flutter (Cardiac disorders) | 2 (2)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Atrioventricular block (Cardiac disorders) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 4 (4)
Atrioventricular block second degree (Cardiac disorders) | 2 (2)
Bradyarrhythmia (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 3 (3)
Cardiac arrest (Cardiac disorders) | 8 (8)
Cardiac failure (Cardiac disorders) | 28 (32)
Cardiac failure acute (Cardiac disorders) | 2 (2)
Cardiac failure chronic (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 14 (14)
Cardiac ventricular thrombosis (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Cardiomegaly (Cardiac disorders) | 1 (1)
Cor pulmonale (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 9 (10)
Coronary artery stenosis (Cardiac disorders) | 2 (2)
Hypertensive heart disease (Cardiac disorders) | 2 (2)
Ischaemic cardiomyopathy (Cardiac disorders) | 2 (2)
Mitral valve incompetence (Cardiac disorders) | 2 (2)
Mitral valve stenosis (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 18 (18)
Myocardial ischaemia (Cardiac disorders) | 8 (8)
Myocarditis (Cardiac disorders) | 1 (1)
Nodal rhythm (Cardiac disorders) | 1 (1)
Parasystole (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (2)
Pericarditis (Cardiac disorders) | 1 (1)
Prinzmetal angina (Cardiac disorders) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 3 (3)
Supraventricular tachycardia (Cardiac disorders) | 2 (2)
Tachyarrhythmia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Left ventricle outflow tract obstruction (Congenital, familial and genetic disorders) | 1 (1)
Type v hyperlipidaemia (Congenital, familial and genetic disorders) | 1 (1)
Acute vestibular syndrome (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 3 (3)
Vertigo positional (Ear and labyrinth disorders) | 1 (1)
Goitre (Endocrine disorders) | 2 (2)
Toxic goitre (Endocrine disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Cataract nuclear (Eye disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Macular hole (Eye disorders) | 1 (1)
Retinal artery occlusion (Eye disorders) | 1 (1)
Retinal detachment (Eye disorders) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 7 (7)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 8 (8)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 4 (4)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 8 (8)
Intestinal obstruction (Gastrointestinal disorders) | 5 (5)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1)
Mallory-weiss syndrome (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Obstructive pancreatitis (Gastrointestinal disorders) | 3 (3)
Oesophageal perforation (Gastrointestinal disorders) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 2 (2)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1)
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (3)
Spigelian hernia (Gastrointestinal disorders) | 1 (1)
Tooth impacted (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3)
Volvulus (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Accidental death (General disorders) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Chest pain (General disorders) | 8 (8)
Death (General disorders) | 6 (6)
General physical health deterioration (General disorders) | 2 (2)
Multiple organ dysfunction syndrome (General disorders) | 3 (3)
Oedema (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 2 (2)
Pyrexia (General disorders) | 3 (3)
Sudden death (General disorders) | 1 (1)
Vascular stent stenosis (General disorders) | 1 (1)
Vascular stent thrombosis (General disorders) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 2 (2)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 5 (5)
Cholecystitis acute (Hepatobiliary disorders) | 4 (4)
Cholelithiasis (Hepatobiliary disorders) | 5 (5)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1)
Hepatic haematoma (Hepatobiliary disorders) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1)
Abscess (Infections and infestations) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1)
Appendicitis (Infections and infestations) | 5 (5)
Appendicitis perforated (Infections and infestations) | 2 (2)
Arthritis bacterial (Infections and infestations) | 1 (1)
Atypical pneumonia (Infections and infestations) | 1 (1)
Bacterial infection (Infections and infestations) | 2 (2)
Bone tuberculosis (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 6 (6)
Cellulitis (Infections and infestations) | 8 (9)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Cytomegalovirus colitis (Infections and infestations) | 1 (1)
Diabetic foot infection (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 7 (7)
Endophthalmitis (Infections and infestations) | 2 (2)
Erysipelas (Infections and infestations) | 4 (4)
Escherichia bacteraemia (Infections and infestations) | 1 (1)
Escherichia infection (Infections and infestations) | 1 (1)
Escherichia pyelonephritis (Infections and infestations) | 1 (1)
Gastric ulcer helicobacter (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (3)
Herpes simplex (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 2 (2)
Infectious pleural effusion (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 9 (9)
Joint abscess (Infections and infestations) | 1 (1)
Liver abscess (Infections and infestations) | 2 (2)
Localised infection (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 3 (4)
Necrotising fasciitis (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1)
Paraoesophageal abscess (Infections and infestations) | 1 (1)
Pathogen resistance (Infections and infestations) | 1 (1)
Peritonitis (Infections and infestations) | 4 (4)
Peritonsillar abscess (Infections and infestations) | 1 (1)
Pilonidal cyst (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 54 (58)
Pneumonia haemophilus (Infections and infestations) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 4 (4)
Respiratory tract infection (Infections and infestations) | 4 (6)
Respiratory tract infection bacterial (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 10 (10)
Septic shock (Infections and infestations) | 2 (4)
Systemic candida (Infections and infestations) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 17 (17)
Urosepsis (Infections and infestations) | 1 (1)
Vulval abscess (Infections and infestations) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 2 (3)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 4 (4)
Cardiac valve rupture (Injury, poisoning and procedural complications) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 4 (4)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 5 (5)
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 (3)
Femur fracture (Injury, poisoning and procedural complications) | 8 (8)
Head injury (Injury, poisoning and procedural complications) | 6 (6)
Hip fracture (Injury, poisoning and procedural complications) | 3 (3)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Kidney contusion (Injury, poisoning and procedural complications) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 2 (2)
Liver contusion (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 3 (3)
Multiple injuries (Injury, poisoning and procedural complications) | 2 (2)
Patella fracture (Injury, poisoning and procedural complications) | 2 (2)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1)
Poisoning (Injury, poisoning and procedural complications) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Post procedural swelling (Injury, poisoning and procedural complications) | 1 (1)
Pulmonary contusion (Injury, poisoning and procedural complications) | 3 (3)
Radiation proctitis (Injury, poisoning and procedural complications) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 5 (5)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Shunt occlusion (Injury, poisoning and procedural complications) | 1 (1)
Skin injury (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 5 (5)
Spinal column injury (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 5 (5)
Subdural haematoma (Injury, poisoning and procedural complications) | 7 (7)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 3 (3)
Transfusion-related acute lung injury (Injury, poisoning and procedural complications) | 1 (1)
Traumatic liver injury (Injury, poisoning and procedural complications) | 1 (1)
Ulnar nerve injury (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 3 (3)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Viith nerve injury (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 2 (2)
Blood potassium decreased (Investigations) | 1 (1)
Blood pressure increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 (2)
Gout (Metabolism and nutrition disorders) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (5)
Latent autoimmune diabetes in adults (Metabolism and nutrition disorders) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 2 (3)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 (4)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 15 (16)
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 3 (3)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (2)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 (1)
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
B precursor type acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (12)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ganglioneuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hypopharyngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Insulinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Marginal zone lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Ovarian cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Penile cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Renal cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Basal ganglia haemorrhage (Nervous system disorders) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 2 (2)
Carotid sinus syndrome (Nervous system disorders) | 1 (1)
Cerebellar ataxia (Nervous system disorders) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 2 (2)
Cerebral haemorrhage (Nervous system disorders) | 4 (4)
Cerebral infarction (Nervous system disorders) | 8 (9)
Cerebral ischaemia (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 14 (14)
Coma (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4)
Embolic cerebral infarction (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Facial paralysis (Nervous system disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 2 (2)
Haemorrhagic stroke (Nervous system disorders) | 1 (1)
Haemorrhagic transformation stroke (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 4 (4)
Lacunar stroke (Nervous system disorders) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1)
Myoclonus (Nervous system disorders) | 1 (1)
Neuroglycopenia (Nervous system disorders) | 1 (1)
Normal pressure hydrocephalus (Nervous system disorders) | 1 (1)
Petit mal epilepsy (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Radicular pain (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 3 (3)
Syncope (Nervous system disorders) | 8 (8)
Transient global amnesia (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 11 (11)
Vith nerve paralysis (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 3 (3)
Depression (Psychiatric disorders) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 6 (6)
Bladder obstruction (Renal and urinary disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 6 (6)
End stage renal disease (Renal and urinary disorders) | 1 (1)
Glomerulonephritis (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 4 (4)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Prerenal failure (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 4 (4)
Renal impairment (Renal and urinary disorders) | 1 (1)
Renal injury (Renal and urinary disorders) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 3 (3)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 3 (3)
Prostatitis (Reproductive system and breast disorders) | 1 (1)
Rectocele (Reproductive system and breast disorders) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Sinus perforation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Aortic aneurysm (Vascular disorders) | 3 (3)
Aortic dissection (Vascular disorders) | 1 (1)
Aortic rupture (Vascular disorders) | 1 (1)
Aortic stenosis (Vascular disorders) | 2 (2)
Arterial rupture (Vascular disorders) | 1 (1)
Arteriosclerosis (Vascular disorders) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Embolism venous (Vascular disorders) | 1 (1)
Extremity necrosis (Vascular disorders) | 2 (2)
Haematoma (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 10 (10)
Hypertensive crisis (Vascular disorders) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 1 (1)
Intermittent claudication (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 3 (3)
Peripheral venous disease (Vascular disorders) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1)
Poor peripheral circulation (Vascular disorders) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1)
Subclavian steal syndrome (Vascular disorders) | 1 (1)
Temporal arteritis (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Senile dementia (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HZ/su Group (N=8687)
Anaemia (Blood and lymphatic system disorders) | 4 (4)
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 3 (4)
Pseudolymphoma (Blood and lymphatic system disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 2 (2)
Arrhythmia (Cardiac disorders) | 9 (11)
Atrial fibrillation (Cardiac disorders) | 11 (11)
Atrioventricular block (Cardiac disorders) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Cardiovascular disorder (Cardiac disorders) | 1 (1)
Chronic left ventricular failure (Cardiac disorders) | 1 (1)
Dilatation ventricular (Cardiac disorders) | 1 (1)
Extrasystoles (Cardiac disorders) | 1 (1)
Hypertensive heart disease (Cardiac disorders) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1)
Mitral valve prolapse (Cardiac disorders) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 2 (2)
Palpitations (Cardiac disorders) | 10 (11)
Pericardial effusion (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 2 (2)
Cerumen impaction (Ear and labyrinth disorders) | 3 (3)
Deafness (Ear and labyrinth disorders) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 12 (12)
Ear pruritus (Ear and labyrinth disorders) | 1 (1)
Excessive cerumen production (Ear and labyrinth disorders) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 3 (3)
Meniere's disease (Ear and labyrinth disorders) | 1 (1)
Motion sickness (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 5 (6)
Vertigo (Ear and labyrinth disorders) | 18 (20)
Vertigo positional (Ear and labyrinth disorders) | 2 (2)
Hyperparathyroidism secondary (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 3 (3)
Accommodation disorder (Eye disorders) | 1 (1)
Age-related macular degeneration (Eye disorders) | 1 (1)
Angle closure glaucoma (Eye disorders) | 1 (1)
Asthenopia (Eye disorders) | 1 (1)
Blepharitis (Eye disorders) | 4 (4)
Blepharospasm (Eye disorders) | 1 (1)
Blindness transient (Eye disorders) | 1 (1)
Cataract (Eye disorders) | 3 (3)
Conjunctival haemorrhage (Eye disorders) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 3 (3)
Dry eye (Eye disorders) | 4 (4)
Eye haematoma (Eye disorders) | 1 (1)
Eye haemorrhage (Eye disorders) | 3 (3)
Eye inflammation (Eye disorders) | 1 (1)
Eye irritation (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 8 (9)
Eye swelling (Eye disorders) | 3 (3)
Glaucoma (Eye disorders) | 1 (1)
Iridocyclitis (Eye disorders) | 1 (1)
Lacrimation decreased (Eye disorders) | 4 (4)
Lacrimation increased (Eye disorders) | 2 (3)
Ocular discomfort (Eye disorders) | 1 (1)
Ocular hyperaemia (Eye disorders) | 1 (1)
Panophthalmitis (Eye disorders) | 1 (1)
Photophobia (Eye disorders) | 2 (2)
Retinal disorder (Eye disorders) | 1 (1)
Retinal drusen (Eye disorders) | 1 (1)
Retinal haemorrhage (Eye disorders) | 1 (1)
Retinal vein occlusion (Eye disorders) | 1 (1)
Swelling of eyelid (Eye disorders) | 2 (2)
Ulcerative keratitis (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 10 (11)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 14 (15)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 39 (45)
Anal inflammation (Gastrointestinal disorders) | 1 (1)
Angular cheilitis (Gastrointestinal disorders) | 1 (1)
Anorectal discomfort (Gastrointestinal disorders) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 26 (26)
Crohn's disease (Gastrointestinal disorders) | 1 (1)
Dental caries (Gastrointestinal disorders) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 107 (114)
Diverticulum (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 8 (9)
Dyspepsia (Gastrointestinal disorders) | 19 (20)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Enteritis (Gastrointestinal disorders) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 3 (3)
Eructation (Gastrointestinal disorders) | 2 (2)
Faeces soft (Gastrointestinal disorders) | 2 (2)
Flatulence (Gastrointestinal disorders) | 4 (4)
Food poisoning (Gastrointestinal disorders) | 1 (1)
Gastric disorder (Gastrointestinal disorders) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 8 (9)
Gastritis erosive (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 3 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 12 (12)
Gingival bleeding (Gastrointestinal disorders) | 1 (1)
Gingival ulceration (Gastrointestinal disorders) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 4 (4)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1)
Lip pain (Gastrointestinal disorders) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 3 (3)
Lip ulceration (Gastrointestinal disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 6 (6)
Nausea (Gastrointestinal disorders) | 164 (184)
Odynophagia (Gastrointestinal disorders) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1)
Oral discomfort (Gastrointestinal disorders) | 1 (2)
Oral mucosal blistering (Gastrointestinal disorders) | 2 (2)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Paraesthesia oral (Gastrointestinal disorders) | 2 (3)
Peptic ulcer (Gastrointestinal disorders) | 2 (2)
Periodontal disease (Gastrointestinal disorders) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Rectal tenesmus (Gastrointestinal disorders) | 1 (1)
Reflux gastritis (Gastrointestinal disorders) | 1 (1)
Retching (Gastrointestinal disorders) | 1 (1)
Salivary gland calculus (Gastrointestinal disorders) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Tongue blistering (Gastrointestinal disorders) | 1 (1)
Tongue dry (Gastrointestinal disorders) | 1 (1)
Tongue ulceration (Gastrointestinal disorders) | 1 (1)
Tooth disorder (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 14 (14)
Vomiting (Gastrointestinal disorders) | 37 (38)
Administration site discomfort (General disorders) | 1 (1)
Administration site erythema (General disorders) | 20 (21)
Administration site oedema (General disorders) | 1 (1)
Administration site pain (General disorders) | 50 (57)
Administration site pruritus (General disorders) | 4 (4)
Administration site swelling (General disorders) | 13 (13)
Administration site warmth (General disorders) | 1 (1)
Application site burn (General disorders) | 2 (2)
Asthenia (General disorders) | 74 (81)
Axillary pain (General disorders) | 3 (3)
Chest discomfort (General disorders) | 4 (4)
Chest pain (General disorders) | 13 (14)
Chills (General disorders) | 319 (366)
Cyst (General disorders) | 1 (1)
Discomfort (General disorders) | 15 (16)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 384 (448)
Feeling abnormal (General disorders) | 7 (7)
Feeling cold (General disorders) | 47 (52)
Feeling hot (General disorders) | 29 (31)
General physical health deterioration (General disorders) | 7 (7)
Hyperthermia (General disorders) | 2 (2)
Inflammation (General disorders) | 2 (2)
Influenza like illness (General disorders) | 65 (74)
Injection site bruising (General disorders) | 14 (14)
Injection site discomfort (General disorders) | 13 (14)
Injection site eczema (General disorders) | 3 (3)
Injection site erythema (General disorders) | 1311 (1717)
Injection site exfoliation (General disorders) | 1 (1)
Injection site extravasation (General disorders) | 1 (1)
Injection site haematoma (General disorders) | 13 (13)
Injection site haemorrhage (General disorders) | 5 (5)
Injection site hyperaesthesia (General disorders) | 7 (8)
Injection site hypersensitivity (General disorders) | 3 (3)
Injection site hypertrophy (General disorders) | 1 (1)
Injection site hypoaesthesia (General disorders) | 9 (9)
Injection site induration (General disorders) | 64 (73)
Injection site inflammation (General disorders) | 85 (94)
Injection site irritation (General disorders) | 4 (4)
Injection site joint discomfort (General disorders) | 1 (2)
Injection site joint pain (General disorders) | 24 (25)
Injection site mass (General disorders) | 6 (7)
Injection site movement impairment (General disorders) | 13 (13)
Injection site nodule (General disorders) | 1 (1)
Injection site oedema (General disorders) | 23 (24)
Injection site pain (General disorders) | 3173 (4579)
Injection site paraesthesia (General disorders) | 6 (6)
Injection site pruritus (General disorders) | 248 (299)
Injection site rash (General disorders) | 46 (51)
Injection site reaction (General disorders) | 24 (27)
Injection site scab (General disorders) | 1 (1)
Injection site swelling (General disorders) | 928 (1194)
Injection site urticaria (General disorders) | 4 (4)
Injection site vesicles (General disorders) | 1 (1)
Injection site warmth (General disorders) | 177 (211)
Malaise (General disorders) | 226 (258)
Nodule (General disorders) | 2 (2)
Oedema peripheral (General disorders) | 10 (10)
Pain (General disorders) | 183 (213)
Peripheral swelling (General disorders) | 15 (16)
Polyp (General disorders) | 1 (1)
Pyrexia (General disorders) | 1038 (1261)
Sluggishness (General disorders) | 1 (1)
Swelling (General disorders) | 2 (2)
Temperature intolerance (General disorders) | 1 (1)
Temperature regulation disorder (General disorders) | 7 (8)
Tenderness (General disorders) | 1 (1)
Thirst (General disorders) | 2 (2)
Vaccination site erythema (General disorders) | 51 (58)
Vaccination site induration (General disorders) | 3 (3)
Vaccination site inflammation (General disorders) | 2 (2)
Vaccination site irritation (General disorders) | 2 (2)
Vaccination site mass (General disorders) | 1 (1)
Vaccination site oedema (General disorders) | 8 (8)
Vaccination site pain (General disorders) | 135 (156)
Vaccination site paraesthesia (General disorders) | 1 (1)
Vaccination site pruritus (General disorders) | 11 (12)
Vaccination site rash (General disorders) | 1 (2)
Vaccination site swelling (General disorders) | 37 (40)
Vaccination site warmth (General disorders) | 7 (7)
Vessel puncture site bruise (General disorders) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 3 (3)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1)
Allergy to animal (Immune system disorders) | 1 (1)
Allergy to arthropod bite (Immune system disorders) | 1 (1)
Food allergy (Immune system disorders) | 2 (2)
Hypersensitivity (Immune system disorders) | 6 (6)
Multiple allergies (Immune system disorders) | 1 (1)
Reaction to food additive (Immune system disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 4 (4)
Abscess (Infections and infestations) | 1 (1)
Acarodermatitis (Infections and infestations) | 1 (1)
Acute sinusitis (Infections and infestations) | 3 (3)
Blastocystis infection (Infections and infestations) | 1 (1)
Borrelia infection (Infections and infestations) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 40 (41)
Cellulitis (Infections and infestations) | 8 (8)
Chronic sinusitis (Infections and infestations) | 1 (1)
Conjunctivitis (Infections and infestations) | 18 (18)
Cystitis (Infections and infestations) | 17 (17)
Dacryocystitis (Infections and infestations) | 1 (1)
Dengue fever (Infections and infestations) | 1 (1)
Dermatophytosis of nail (Infections and infestations) | 2 (2)
Diverticulitis (Infections and infestations) | 2 (2)
Ear infection (Infections and infestations) | 6 (6)
Erysipelas (Infections and infestations) | 5 (5)
Eye infection (Infections and infestations) | 4 (4)
Folliculitis (Infections and infestations) | 3 (3)
Fungal infection (Infections and infestations) | 1 (1)
Fungal skin infection (Infections and infestations) | 2 (2)
Furuncle (Infections and infestations) | 2 (2)
Gastric infection (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 17 (17)
Gastroenteritis viral (Infections and infestations) | 2 (2)
Gastrointestinal viral infection (Infections and infestations) | 1 (1)
Genital herpes (Infections and infestations) | 1 (1)
Gingivitis (Infections and infestations) | 6 (6)
Helicobacter infection (Infections and infestations) | 1 (1)
Herpes simplex (Infections and infestations) | 19 (22)
Hordeolum (Infections and infestations) | 5 (5)
Impetigo (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 52 (54)
Injection site cellulitis (Infections and infestations) | 2 (2)
Injection site infection (Infections and infestations) | 2 (2)
Labyrinthitis (Infections and infestations) | 1 (1)
Localised infection (Infections and infestations) | 5 (5)
Lower respiratory tract infection (Infections and infestations) | 21 (21)
Lyme disease (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 228 (239)
Onychomycosis (Infections and infestations) | 5 (5)
Oral candidiasis (Infections and infestations) | 4 (4)
Oral fungal infection (Infections and infestations) | 1 (1)
Oral herpes (Infections and infestations) | 31 (34)
Oral infection (Infections and infestations) | 1 (1)
Otitis externa (Infections and infestations) | 2 (2)
Otitis media (Infections and infestations) | 3 (3)
Pathogen resistance (Infections and infestations) | 1 (1)
Periodontitis (Infections and infestations) | 5 (5)
Pertussis (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 16 (16)
Pharyngotonsillitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 6 (6)
Pulpitis dental (Infections and infestations) | 2 (2)
Pyelonephritis (Infections and infestations) | 2 (2)
Respiratory tract infection (Infections and infestations) | 13 (13)
Respiratory tract infection viral (Infections and infestations) | 3 (3)
Rhinitis (Infections and infestations) | 18 (18)
Sinusitis (Infections and infestations) | 25 (26)
Skin candida (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 3 (3)
Subcutaneous abscess (Infections and infestations) | 1 (1)
Syphilis (Infections and infestations) | 1 (1)
Testicular abscess (Infections and infestations) | 1 (1)
Tinea infection (Infections and infestations) | 1 (1)
Tinea pedis (Infections and infestations) | 6 (7)
Tongue fungal infection (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 5 (5)
Tooth abscess (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 4 (4)
Tracheitis (Infections and infestations) | 3 (4)
Tracheobronchitis (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 80 (86)
Urinary tract infection (Infections and infestations) | 63 (66)
Vaginal infection (Infections and infestations) | 2 (2)
Vaginitis gardnerella (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 6 (6)
Viral upper respiratory tract infection (Infections and infestations) | 3 (3)
Zika virus infection (Infections and infestations) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (2)
Animal bite (Injury, poisoning and procedural complications) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 8 (8)
Arthropod sting (Injury, poisoning and procedural complications) | 2 (2)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 11 (11)
Deafness traumatic (Injury, poisoning and procedural complications) | 1 (1)
Ear injury (Injury, poisoning and procedural complications) | 2 (2)
Epicondylitis (Injury, poisoning and procedural complications) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 11 (12)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 5 (5)
Heat stroke (Injury, poisoning and procedural complications) | 2 (2)
Joint injury (Injury, poisoning and procedural complications) | 5 (5)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 5 (5)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 4 (4)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1)
Skin injury (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 4 (4)
Snake bite (Injury, poisoning and procedural complications) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (2)
Splinter (Injury, poisoning and procedural complications) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (2)
Tooth fracture (Injury, poisoning and procedural complications) | 3 (3)
Tooth injury (Injury, poisoning and procedural complications) | 1 (1)
Traumatic arthritis (Injury, poisoning and procedural complications) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 2 (2)
Wrist fracture (Injury, poisoning and procedural complications) | 3 (3)
Blood cholesterol increased (Investigations) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1)
Blood iron decreased (Investigations) | 1 (1)
Blood pressure decreased (Investigations) | 1 (1)
Blood pressure diastolic increased (Investigations) | 1 (1)
Blood pressure increased (Investigations) | 3 (3)
Blood triglycerides increased (Investigations) | 1 (1)
Blood urea decreased (Investigations) | 1 (1)
Blood uric acid increased (Investigations) | 1 (1)
Body temperature increased (Investigations) | 76 (86)
Cardiac murmur (Investigations) | 3 (3)
Haemoglobin decreased (Investigations) | 1 (1)
Heart rate increased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 15 (15)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Dyslipidaemia (Metabolism and nutrition disorders) | 3 (3)
Gout (Metabolism and nutrition disorders) | 12 (12)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 8 (8)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3)
Hyperlipidaemia (Metabolism and nutrition disorders) | 4 (4)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (4)
Hypovitaminosis (Metabolism and nutrition disorders) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 7 (7)
Vitamin b12 deficiency (Metabolism and nutrition disorders) | 1 (1)
Vitamin d deficiency (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 212 (237)
Arthritis (Musculoskeletal and connective tissue disorders) | 5 (5)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 100 (106)
Bone decalcification (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 13 (14)
Bursitis (Musculoskeletal and connective tissue disorders) | 3 (3)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Foot deformity (Musculoskeletal and connective tissue disorders) | 2 (2)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Growing pains (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc space narrowing (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 2 (3)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 8 (8)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 4 (5)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 24 (30)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 4 (4)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 11 (12)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 53 (55)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 17 (18)
Myalgia (Musculoskeletal and connective tissue disorders) | 386 (481)
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 1 (1)
Myosclerosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 42 (43)
Nuchal rigidity (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 27 (30)
Osteopenia (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 103 (115)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 3 (3)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 4 (4)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 2 (2)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 (2)
Scoliosis (Musculoskeletal and connective tissue disorders) | 3 (3)
Senile osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 2 (2)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 2 (2)
Tendon pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Tendonitis (Musculoskeletal and connective tissue disorders) | 6 (6)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 3 (3)
Torticollis (Musculoskeletal and connective tissue disorders) | 2 (3)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Aphonia (Nervous system disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1)
Burning sensation (Nervous system disorders) | 2 (2)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 2 (2)
Cognitive disorder (Nervous system disorders) | 1 (1)
Dementia alzheimer's type (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 117 (126)
Dysgeusia (Nervous system disorders) | 3 (3)
Essential tremor (Nervous system disorders) | 1 (1)
Facial paralysis (Nervous system disorders) | 1 (1)
Hand-arm vibration syndrome (Nervous system disorders) | 1 (1)
Head discomfort (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 678 (896)
Hyperaesthesia (Nervous system disorders) | 2 (2)
Hypersomnia (Nervous system disorders) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 6 (6)
Intercostal neuralgia (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 27 (31)
Loss of consciousness (Nervous system disorders) | 2 (2)
Memory impairment (Nervous system disorders) | 1 (1)
Mental impairment (Nervous system disorders) | 2 (3)
Migraine (Nervous system disorders) | 15 (18)
Morton's neuralgia (Nervous system disorders) | 1 (1)
Muscle contractions involuntary (Nervous system disorders) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 3 (3)
Paraesthesia (Nervous system disorders) | 6 (6)
Poor quality sleep (Nervous system disorders) | 5 (6)
Presyncope (Nervous system disorders) | 2 (2)
Radiculopathy (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 15 (15)
Sensory disturbance (Nervous system disorders) | 1 (1)
Sinus headache (Nervous system disorders) | 2 (2)
Somnolence (Nervous system disorders) | 22 (22)
Syncope (Nervous system disorders) | 6 (6)
Taste disorder (Nervous system disorders) | 1 (1)
Tension headache (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (2)
Tremor (Nervous system disorders) | 13 (13)
Trigeminal neuralgia (Nervous system disorders) | 2 (2)
Vertebral artery occlusion (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 5 (5)
Depressed mood (Psychiatric disorders) | 6 (6)
Depression (Psychiatric disorders) | 4 (4)
Generalised anxiety disorder (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 32 (34)
Irritability (Psychiatric disorders) | 1 (2)
Listless (Psychiatric disorders) | 2 (2)
Middle insomnia (Psychiatric disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 4 (4)
Sleep disorder (Psychiatric disorders) | 6 (6)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Bladder prolapse (Renal and urinary disorders) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 1 (1)
Chromaturia (Renal and urinary disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 3 (3)
Dysuria (Renal and urinary disorders) | 4 (4)
Ketonuria (Renal and urinary disorders) | 1 (1)
Nephroangiosclerosis (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Nocturia (Renal and urinary disorders) | 6 (6)
Pollakiuria (Renal and urinary disorders) | 3 (3)
Polyuria (Renal and urinary disorders) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1)
Renal pain (Renal and urinary disorders) | 1 (1)
Urethral polyp (Renal and urinary disorders) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 3 (3)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1)
Breast cyst (Reproductive system and breast disorders) | 1 (1)
Breast enlargement (Reproductive system and breast disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 2 (2)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 4 (4)
Vulvar erosion (Reproductive system and breast disorders) | 1 (1)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (1)
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 91 (96)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 (13)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 18 (19)
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 52 (57)
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 19 (20)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 2 (2)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 4 (4)
Blister (Skin and subcutaneous tissue disorders) | 8 (8)
Cold sweat (Skin and subcutaneous tissue disorders) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 16 (16)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 5 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 26 (27)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 29 (30)
Generalised erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 22 (23)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Intertrigo (Skin and subcutaneous tissue disorders) | 1 (1)
Macule (Skin and subcutaneous tissue disorders) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 5 (5)
Papule (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 57 (62)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 11 (11)
Psoriasis (Skin and subcutaneous tissue disorders) | 2 (2)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 49 (51)
Rash erythematous (Skin and subcutaneous tissue disorders) | 3 (3)
Rash generalised (Skin and subcutaneous tissue disorders) | 2 (2)
Rash macular (Skin and subcutaneous tissue disorders) | 3 (3)
Rash maculovesicular (Skin and subcutaneous tissue disorders) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 3 (3)
Rash pruritic (Skin and subcutaneous tissue disorders) | 5 (5)
Rosacea (Skin and subcutaneous tissue disorders) | 3 (3)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 3 (3)
Sensitive skin (Skin and subcutaneous tissue disorders) | 1 (1)
Skin fissures (Skin and subcutaneous tissue disorders) | 2 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 3 (3)
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 9 (11)
Urticaria contact (Skin and subcutaneous tissue disorders) | 1 (1)
Vasculitic ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Essential hypertension (Vascular disorders) | 1 (1)
Flushing (Vascular disorders) | 2 (2)
Haematoma (Vascular disorders) | 4 (4)
Hot flush (Vascular disorders) | 6 (6)
Hypertension (Vascular disorders) | 20 (21)
Hypertensive crisis (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Pallor (Vascular disorders) | 1 (1)
Peripheral venous disease (Vascular disorders) | 2 (2)
Thrombophlebitis (Vascular disorders) | 2 (2)
Thrombophlebitis superficial (Vascular disorders) | 2 (2)
Thrombosis (Vascular disorders) | 2 (2)
Varicose vein (Vascular disorders) | 3 (3)
Mouth swelling (Gastrointestinal disorders) | 1 (1)
Injection site joint swelling (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-05-30): https://cdn.clinicaltrials.gov/large-docs/07/NCT02690207/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/07/NCT02690207/SAP_001.pdf